CLINICAL TRIAL: NCT04714099
Title: Topical Cyclosporine A for the Treatment of Dry Eye: A Randomized Clinical Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine

STUDY DESIGN:
Intervention Model Description: This is prospective randomized comparative clinical study that included 80 eyes of 40 patients with moderate to severe DED. Patients were divided into two groups; group A received topical CsA 0.05% for 3 months, and group B were controls.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical CsA (Experimental): Group A received topical CsA 0.05% for 3 months
  Interventions: Drug: Topical Cyclosporine A
- Control (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topical Cyclosporine A — In our study we used 0.05% CsA prepared in castor oil by transferring (20ml ) of sterile castor oil in a sterile glass vial under laminar flow, removing a volume (400ul)of oil with micropipette (sterile tips), and replacing this volume with an equal volume of alcoholic CsA solution [200mg cyclosporine in 8 ml ethanol (96%)] under laminar flow.
  Arms: Topical CsA
Drug: Placebo — Placebo
  Arms: Control

SUMMARY:
Since the initial description, the therapeutic efficacy of CsA for human KCS has been well documented, with evidence ranging from several small single center randomized double-masked clinical trials to several large multicenter randomized, double-masked clinical trials.(10-12) Therefore, the aim of the work is to evaluate the effect of using topical CsA in treatment of moderate to severe dry eye.

DETAILED DESCRIPTION:
Dry eye disease (DED) is known to be among the most frequently occuring ocular morbidities. It is a growing public health concern affecting 25% of patients who visit ophthalmic clinics.For many years, DED was considered to be limited to dryness of the eyes due to decrease in the aqueous phase in the tear film. In 2007, the International Dry Eye Workshop discussed the definition and classification of DED and developed a new vision for the definition and the three-part classification of DED on the basis of etiology, mechanism, and severity of DED. Moreover, DED can be episodic or chronic. Episodic DED occurs when environmental or visual tasks with reduced blinking overwhelm the stability of the tear and produce symptomatic DED. Chronic DED, although aggravated by the same environmental conditions, persists continuously with symptoms and possible damage to the ocular surface. Because the tear film in DED patients is not stable and incapable to maintain the protective qualities that are important for its structure and function, patients usually experience the discomfort manifestations associated with DED such as burning, stinging, foreign body sensation, ocular fatigue, grittiness, tearing, and dryness. Patients may complain of symptoms of DED in the presence or absence of the known signs and DED may be diagnosed based only on the signs observed by a healthcare professional in the absence of symptoms reported by the patients.Since the initial description, the therapeutic efficacy of CsA for human KCS has been well documented, with evidence ranging from several small single center randomized double-masked clinical trials to several large multicenter randomized, double-masked clinical trials.Therefore, the aim of the work is to evaluate the effect of using topical CsA in treatment of moderate to severe dry eye.

ELIGIBILITY:
Inclusion Criteria:

* We included all patients with moderate to severe dry eye disease (grade 3 or grade 4) with the following criteria: The tear film break up time ≤5 seconds for grade 3 and immediate for grade 4, schirmer test with anesthetic is ≤5 millimeters for grade 3 and ≤2 millimeters for grade 4, corneal or conjunctival staining pattern with fluorescein is abnormal and consistent with an abnormal tear film. Oxford grade II or more, meibomian gland dysfunction is documented (inspissation of the meibomian gland orifices, pitting and neovascularization of the eyelid margins) and one or more moderate (≥2+) dry eye related symptoms; including itching, burning, blurred vision, foreign body sensation, photophobia, veiling, and soreness or pain

Exclusion Criteria:

* Exclusion criteria included Post LASIK patients, Post radiation fibrosis of lacrimal gland, Vitamin A deficiency, Conjunctival scarring (advanced trachoma, chemical burn, OCP), Drugs (anti-histaminics, anti-cholinergic, anti-psychotics, selective serotonin uptake inhibitors), Patients with familial dysautonomia (Riley-Day syndrome), Use of systemic or topical CsA in the previous 90 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Tear Break up Time | 3 months
  Measuring the time lapse between last blink after instillation of fluorescein and appearance of the first dry spot on the corneal surface

SECONDARY OUTCOMES:
Schirmer test | 3 months
  It was performed by placing a thin strip of filter paper in the inferior cul-de-sac following the instillation of topical anesthetic; then, the eyes are closed for 5 minutes, and the amount of wetting of the paper strip is measured. Measurement of less than 5mm is abnormal; 5-10 mm is equivocal.
Intra ocular pressure | 3 months
  Intra ocular pressure measurement by applanation tonometery
Fluorescein staining (Oxford Grading Scale) | 3 months
  graded on a scale from 0 = none to 5 = severe by Oxford grading system
OSDI Scores | 3 months
  The OSDI is a valid and reliable instrument for measuring the severity of dry eye disease. Subjects in the study completed the OSDI Questionnaire each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Mossallam, PhD, Principal Investigator — Alexandria Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No